CLINICAL TRIAL: NCT06177626
Title: Use of a New Smartphone Application, iBlink, to Determine Changes in Eyeblink Conditioning From Home Training in Individuals With Spinocerebellar Ataxias
Brief Title: Use of a New Smartphone Application to Determine Changes in Eyeblink Conditioning From Home Training in Individuals With Spinocerebellar Ataxia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Scott Barbuto, Assistant Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAV2412 (Aim 2 and 3)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Spinocerebellar Ataxias
Keywords: Ataxia; Eyeblink Conditioning; Exercise
MeSH Terms: conditions — Spinocerebellar Ataxias; Ataxia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will know that the participant has received balance or aerobic training, but will not be aware of which group the participant belonged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balance Training (Active Comparator): A physical therapist will tailor a home balance training program for each participant based on pre- training capabilities. Participants will be asked to perform exercises five times a week for thirty-minute sessions. Both dynamic and static exercises will be performed in sitting and standing positions. Exercises will start with stabilizing in a challenging static position and progress to dynamic arm and leg movements in the same or modified position. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be required to log their exercise effort in terms of frequency and level of balance challenge.
  Interventions: Behavioral: Balance Training
- Aerobic Training (Experimental): Participants will be given a stationary exercise bike for home use. They will be instructed to use the exercise bike five times a week for thirty-minute sessions. The exercise intensity prescription will be based on the subject's VO2max determined on pre-test day. The exercise program will start at 60% of intensity per session, and then will be increased by steps of 5% intensity every 2 sessions until participants reach 30 minutes of training at 80% intensity. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be instructed to log each training session. Participants will record duration of exercise, perceived exertion, average heart rate, maximum heart rate, and distance.
  Interventions: Behavioral: Aerobic Training

INTERVENTIONS:
Behavioral: Aerobic Training — Aerobic training on stationary bike 5x a week for 30 minutes a day
  Arms: Aerobic Training
Behavioral: Balance Training — Training 5x a week for 30 minutes. Standard of care.
  Arms: Balance Training

SUMMARY:
Spinocerebellar ataxias are a group of disorders that cause severe disability and can be fatal. There are currently no known disease-modifying treatments available for use, and there is a critical need to find treatments that slow disease progression and allow affected individuals to live more functional lives. Aerobic training show promise as a treatment for these diseases, but it is unclear if training induces neuroplastic changes within the damaged cerebellum to enhance motor learning, or if improvements are primarily caused by changes in leg strength, fatigue, and endurance. It is crucial to understand how the training impacts the brain, and particularly the cerebellum, in order to determine the most effective training regimen. To examine the impact of aerobic exercise on the brain, this study proposes using eyeblink conditioning, a form of motor learning that is dependent on the cerebellum. This study will utilize BlinkLab, a newly developed smartphone application, that overcomes the typical barriers of testing eyeblink conditioning by allowing in-home assessments without the need for expensive equipment. The investigators hypothesize that: 1) individuals with spinocerebellar ataxia will have impaired eyeblink conditioning, and 2) aerobic exercise, but not balance training, will improve eyeblink conditioning in this population. If these hypotheses are found to be true, it would further support that aerobic exercise is able to enhance motor learning in individuals with cerebellar damage.

In Aim 1, investigators will test eyeblink conditioning in individuals with ataxias and follow them over time to see if eyeblink conditioning might be a biomarker for cerebellar ataxia disease progression. The investigators will then use these preliminary results to devise a larger study to further validate eyeblink conditioning as a biomarker for ataxia disease progression. Aim 2 will determine the impact of training on eyeblink conditioning. The investigators expect that aerobic training, but not balance training, will enhance eyeblink conditioning in spinocerebellar ataxia. Finally, Aim 3 will explore the use of eyeblink conditioning as a biomarker of neuroplasticity.

DETAILED DESCRIPTION:
Spinocerebellar ataxias are a group of disorders that cause severe disability due to progressive incoordination. With no FDA approved medications, there is a critical need to find effective treatments. The research team has shown that high intensity aerobic training, defined as 30-minute training sessions, 5 times per week at above 80% maximum heart rate, is a potential treatment, causing clinically significant improvements in ataxia symptoms at 6-months compared to home balance training. However, it is unclear whether aerobic training induces neuroplastic changes within the damaged cerebellum, or if improvements are primarily due to increased leg strength and endurance which help compensate for ataxia and balance deficits.

The investigators hypothesize that aerobic training causes improvements for people with spinocerebellar ataxias by inducing neuroplastic changes within the cerebellum whereas balance training does not. The hypothesis is supported by: 1) Research that balance training in individuals with spinocerebellar ataxia causes increased grey matter volume in the premotor cortex, but no statistically significant changes in the cerebellum. 2) Although not verified in humans, aerobic exercise rescues motor coordination deficits in ataxic mice and improvements correlate with restored cerebellar BDNF levels. 3) TrkB, the BDNF receptor, was vital for improved motor function and reduced Purkinje cell degeneration seen in ataxic rats that performed endurance exercise. Thus, this study proposes that aerobic training increases cerebellar BDNF levels which enhances responsivity to neurotransmitters and downregulates GABA-inhibition. This response, in turn, leads to a fertile environment in the cerebellum with one consequence being improved motor learning.

In order to investigate the impact of aerobic training on cerebellar dependent motor learning, this study will use eyeblink conditioning. In this task, individuals learn to blink in response to a conditioned stimulus that is paired with an unconditioned stimulus. Unfortunately, eyeblink conditioning is costly, requires multiple in-person visits to measure learning, and produces data that necessitates extensive programing and data management skills to interpret. To overcome these barriers, the study collaborators recently developed BlinkLab, an application for the smartphone that can test eyeblink conditioning remotely. This application is low cost, straight-forward for participants to use at home, and produces easily interpretable data. Moreover, the research team has shown that BlinkLab can be used to determine changes in eyeblink conditioning due to aerobic training in healthy individuals. Thus, the goal of this pilot study will be to use the BlinkLab application to study the impact of exercise on eyeblink conditioning serving as a proxy for neuroplastic changes within the cerebellum.

Aim 1) To determine if eyeblink conditioning is a useful biomarker for spinocerebellar ataxias. Preliminary work with BlinkLab indicates that individuals with ataxia have deficits in eyeblink conditioning compared to healthy controls. The study will recruit 40 individuals with spinocerebellar ataxia and compare changes in ataxia symptoms to changes in eyeblink conditioning over 6-months. The investigators hypothesize that eyeblink conditioning will worsen as disease progresses.

Aim 2) Impact of aerobic exercise on eyeblink conditioning in spinocerebellar ataxias. Thirty individuals with spinocerebellar ataxias will be randomized to either home balance or aerobic training for 3-months. Participants will undergo eyeblink conditioning using BlinkLab at baseline, 3- and 4-months. Secondary outcome measures will include ataxia severity, leg strength, endurance, fitness, balance, and abilities to do activities of daily living. The investigators hypothesize that individuals in the aerobic group will have improved eyeblink conditioning compared to the balance training group. Furthermore, the investigators expect that improvements in ataxia symptoms will correlate with improvements in eyeblink conditioning.

Exploratory Aim 3) Correlation of eyeblink conditioning changes induced by aerobic training with functional connectivity changes in the cerebellum. Resting state fMRI scans will be taken before and after individuals with spinocerebellar ataxia participate in the 3-month training programs in Aim 2. Investigators will then use the cerebellum as the region of interest to analyze how training impacts functional cerebellar connections. Investigators will explore the relationship between eyeblink conditioning and functional cerebellar changes caused by training to assess the use of eyeblink conditioning as a biomarker of neuroplasticity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spinocerebellar ataxia
* Cerebellar atrophy on MRI
* Prevalence of ataxia on clinical exam (SARA >2)
* Ability to safely ride a stationary exercise bike (SARA sitting sub-score <3)

Exclusion Criteria:

* Parkinson's Disease
* Traumatic Brain Injury
* Stroke
* Alzheimer's Disease
* Heart disease
* Dementia
* Medical instability
* Inability to walk without assistance (SARA gait sub-score >6).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Conditioned Response (CR) Amplitude | 0, 3, and 4 months
  Individual eyelid traces will be normalized by dividing each trace by the maximum signal amplitude of the relevant session. Thus, eyes closed will correspond to a value of 1, and eyes open to a value of 0. A mean baseline Conditioned Response (CR) amplitude will be determined for each participant using the pre-block Conditioned Stimulus (CS) only trials. CR amplitude will then be determined as the maximum signal amplitude value at 430ms, for paired and CS only trials, minus the baseline CR amplitude.

SECONDARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | 0, 3, and 4 months
  SARA is a validated clinical measure of ataxia severity. Scores range from 0 to 40 with higher scores indicating more ataxia symptoms. Each SARA test will be recorded and the order scrambled to blind researchers to time of testing. This test has a sensitivity of 0.99 and specificity of 0.96. Interrater reliability, test-retest reliability, and internal consistency was also determined to be high. SARAhome is a validated home measurement of ataxia symptoms with the participants recording 5 tasks (gait, stance, speech, nose-finger test, and fast alternating hand movements) with a smartphone. Scores range from 0 to 28 with higher scores indicating more ataxia symptoms. SARAhome and the conventional SARA were shown to be highly correlated, and this measurement was deemed reliable for home monitoring of ataxia symptoms. Scores will be used to correlate with changes in eyeblink conditioning in Aim 1.
PROM of Ataxia Score | 0, 3, and 4 months
  The Patient Reported Outcome Measure (PROM) of Ataxia is a 70-item survey that is scored by participants on a 0-4 Likert scale. It asks participants to rate motor domains of gait, lower and upper extremity control, manual dexterity, visual motor control, dysphagia, bowel and bladder function, sleep, fatigue, vertigo, libido, neuropathy, ability to do household chores, driving, self-care, mood, anxiety, motivation, and social interactions. Scores will be used to correlate with changes in eyeblink conditioning as a result of training. Scores range from 0-280 with a higher score indicating a worse outcome.
Quantitative Muscle Testing (QMT) | 0, 3, and 4 months
  QMT has been shown to have excellent intra-rater and inter-rater reliability for the measurement of leg strength. Knee extensor and flexor strength will be determined by measuring maximal voluntary isometric contraction using QMT (Aeverl Medical, Gainesville, GA). This system consists of an adjustable strap, attaching the legs to interface force transducers. Subjects will be tested on an adjustable examination table that anchors the transducer. The generated force is transmitted to an electronic strain-gauge tensiometer and is then recorded and amplified by the data computer-assisted analog to digital acquisition system.
6-minute Walk Test (6MWT) | 0, 3, and 4 months
  The 6MWT is a validated measure of endurance. Individuals will be instructed to walk as far as they can on a 30-meter walkway. It was deemed to have excellent reliability.
Balance Measures | 0, 3, and 4 months
  To monitor balance, the Timed Up and Go (TUG) test will be performed according to standard protocols. Participants will also perform the Dynamic Gait Index (DGI) using the established protocol. Scores on the DGI range from 0 to 24 with lower scores indicating more severe problems with balance and increased risk of falling. Although not determined on individuals with spinocerebellar ataxia, a minimal clinically important difference of 1.9 points was determined for community-dwelling older adults.
Maximal Oxygen Consumption (VO2Max) | 0, 3, and 4 months
  Results from CPET at initial testing will be used to develop training programs for those randomized to the aerobic group. It will also be used as a secondary outcome for Aim 2. Maximal oxygen consumption (VO2max) will be determined by a breath-by-breath measurement of VO2 with a Vmax Encore Metabolic System, while participants perform a progressive ramped exercise test using an electronic-braked lower body cycle ergometer (CareFusion Corp, San Diego, CA).
Maximal Oxygen Consumption (VO2Max) | 0 and 3 months
  Resting State Functional MRI: This measure will be a primary outcome for Aim 3. The anatomical and functional data will be pre-processed and analyzed using Statistical Parametric Mapping (SPM12) and the CONN toolbox Version 14p. Functional data will be pre-processed using a slice scan time correction, realignment (motion correction), registration to structural images and spatial normalization to Montreal Neurological Institute (MNI) standardized space, smoothing with a Gaussian filter of 5.0 mm spatial full width at half maximum value. A conventional band-pass filter over a low-frequency window of interest (0.008-0.09) will also be applied to the resting-state time series. After these preprocessing steps, we will extract signal to noise from the white matter and cerebrospinal fluid by principal component analysis without affecting intrinsic functional connectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University/New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No